CLINICAL TRIAL: NCT06530394
Title: Effects of Increased Greek Yogurt Consumption on Circulating Markers of Bone Metabolism and Inflammation in Senior Adults
Brief Title: Effects of Increased Greek Yogurt Consumption in Senior Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brock University (Other)
Responsible Party: Principal Investigator, Panagiota Klentrou, Professor, Brock University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: REB 23-354
Record Dates: First submitted 2024-07-28; First posted 2024-07-31 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Osteoporosis; Inflammation
MeSH Terms: conditions — Osteoporosis; Inflammation

STUDY DESIGN:
Intervention Model Description: Participants will be invited to participate in this 8-week study, with senior fit participants being randomly assigned into the control (NYEX) or the intervention exercising (GYEX) group and non-senior fit citizens from the Niagara community will be assigned to the intervention non-exercising group (GYNE).
Who Masked: Outcomes Assessor
Masking Description: Independent blind researchers will analyze blood and data using masked participant codes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Greek yogurt exercising group (GYEX) (Experimental): Participants will be asked to consume 2 servings/day (preferably morning and night) of 175 g commercially available GY (0% MF, flavoured, 130 calories, 17 g protein, 225 g calcium (e.g., OIKOS High Protein GY) for a total of 8 weeks. For their convenience, the participants will be provided with appropriate scoops to measure out 175 g of GY per serving of the larger 650 g commercially available, pre-packaged containers. Although it is recommended to consume the two servings morning and night, to increase ecological validity and strengthen the feasibility of the intervention, the timing of the servings will be flexible to facilitate daily routines and lifestyles. For the same reasons, the participants will be able to choose the flavour of their GY.
  Interventions: Dietary Supplement: Greek yogurt
- Control exercising group (NYEX) (No Intervention): During the 8-weeks, participants will be instructed to follow their typical, habitual diet and exercise regimen.
- Intervention non-exercising group (GYNE) (Active Comparator): Participants will be instructed to follow their typical habitual diet. Participants will be asked to consume 2 servings/day (preferably morning and night) of 175 g commercially available GY (0% MF, flavoured, 130 calories, 17 g protein, 225 g calcium; e.g., OIKOS High Protein GY) for a total of 8 weeks. For their convenience, the participants will be provided with appropriate scoops to measure out 175 g of GY per serving of the larger 650 g commercially available, pre-packaged containers. Although it is recommended to consume the two servings morning and night, to increase ecological validity and strengthen the intervention's feasibility, the servings' timing will be flexible to facilitate daily routines and lifestyles. For the same reasons, the participants will be able to choose the flavour of their GY.
  Interventions: Dietary Supplement: Greek yogurt

INTERVENTIONS:
Dietary Supplement: Greek yogurt — Whole food dairy products, such as Greek yogurt (GY), offer a high quality, nutrient-dense snack, high in bone-supporting ingredients, including protein, calcium, and phosphorus. These nutrients are crucial to the structural integrity and strength of bone, i.e., the collagen and hydroxyapatite matrices.
  Arms: Greek yogurt exercising group (GYEX); Intervention non-exercising group (GYNE)

SUMMARY:
This study aims to examine whether Greek yogurt (GY) consumption will lead to beneficial changes in bone metabolism and inflammation, in senior adults, male and female, when combined with regular exercise (senior fit classes; GYEX) and without exercise (GYNE). It is hypothesized that compared to a control group (senior fit classes, no GY; NYEX), an 8-week GY consumption intervention in senior adults with and without exercise will lead to positive effects on body composition, and markers of bone metabolism and inflammation such that the anabolic and anti-inflammatory markers of these physiological processes will increase more than any training-induced catabolic and pro-inflammatory markers (i.e., more than measures observed in the NYNE group).

DETAILED DESCRIPTION:
Participants

The proposed project will follow a randomized controlled parallel design over 8 weeks. A total of 60 senior adults (aged 55+ years; males and females) from the Brock Senior Fit program and Niagara area. All participants will provide written informed consent in order to be included in the study. Potential participants will complete a standardized Get Active screening questionnaire of the Canadian Society for Exercise Physiology. Participants will be excluded from the study if they are injured and unable to participate in classes, have an allergy to dairy foods/dairy protein or have been diagnosed with lactose intolerance.

Study Design and Procedures

Participants will be invited to participate in this 8-week study, with senior fit participants being randomly assigned into the control (NYEX) or the intervention exercising (GYEX) group and non-senior fit citizens from the Niagara community will be assigned to the intervention non-exercising group (GYNE).

Control (NYEX) Group: During the 8-weeks, participants will be instructed to follow their typical, habitual diet and exercise regimen.

Intervention Exercising (GYEX) Group: During the 8 weeks, participants will be instructed to follow their typical, habitual diet and exercise regimen. Participants will be asked to consume 2 servings/day (preferably morning and night) of 175 grams of commercially available GY (0% fat, flavoured, 130 calories, 17 grams protein, 225 grams calcium (e.g., OIKOS High Protein GY) for a total of 8 weeks. For their convenience, the participants will be provided with appropriate scoops to measure out 175 grams of GY per serving of the larger 650-gram commercially available, pre-packaged containers. Although it is recommended to consume the two servings morning and night, to increase ecological validity and strengthen the feasibility of the intervention, the timing of the servings will be flexible to facilitate daily routines and lifestyles. For the same reasons, the participants will be able to choose the flavour of their GY.

Intervention Non-Exercising (GYNE) Group: During the 8-weeks participants will be instructed to follow their typical habitual diet. Participants will be asked to consume 2 servings/day (preferably morning and night) of 175 grams of commercially available GY (0% fat, flavoured, 130 calories, 17 grams protein, 225 grams calcium; e.g., OIKOS High Protein GY) for a total of 8 weeks. For their convenience, the participants will be provided with appropriate scoops to measure out 175 grams of GY per serving of the larger 650-gram commercially available, pre-packaged containers. Although it is recommended to consume the two servings morning and night, to increase ecological validity and strengthen the feasibility of the intervention, the timing of the servings will be flexible to facilitate daily routines and lifestyles. For the same reasons, the participants will be able to choose the flavour of their GY.

At weeks 0 and 8 (the beginning and end of the study), all participants will complete a series of nutrition and activity questionnaires and have their body composition measured, and their fasted, resting morning blood collected. All participants will be instructed not to consume any food or liquids (except water, as needed) 8 hours before the time of their blood draw, not to exercise for 12 hours before the blood draw, and not to make any changes to their normal routines. These measurements will take place in the Applied Physiology Laboratory at Brock University by the same investigators.

Measurements

The following measurements will be collected at the beginning (week 0) and completion of the study (week 8).

Blood analysis: A total of 10 microliters (mL) of blood will be collected from an antecubital vein by a certified phlebotomist or registered nurse using a standardized venipuncture technique. All blood samples will be centrifuged for 10 minutes. Serum and plasma will be aliquoted into pre-labelled Eppendorf tubes and stored at -80°C until analysis. The serum concentrations of markers and regulators of bone remodelling will be analyzed in duplicate using ELISA kits for osteocalcin, amino-terminal propeptide of type I collagen (P1NP), and osteoprotegerin (OPG)) and bone resorption (C-telopeptides of type I collagen (CTX), sclerostin, receptor activator of nuclear factor kappa-Β ligand (RANKL), and parathyroid hormone (PTH). The plasma concentrations of inflammatory cytokines, including interleukin-6 (IL6), interleukin-10 (IL10), tumour necrosis factor-alpha (TNFα), insulin-like growth factor 1 (IGF1), irisin and brain-derived neurotrophic factor (BDNF), will be measured in triplicate using commercially available ELLA kits. Plasma analyses will be performed in-house at the Centre for Bone and Muscle Health at Brock University.

Body Composition: Body mass and body composition, including lean body mass (LBM), fat mass (FM), and relative body fat percent (%BF), will be measured using bioelectrical impedance analysis (BIA; InBody520 bioelectrical impedance analysis system (Biospace Co. Inc. Los Angeles, CA, USA) following standard procedures.

Dietary and Physical Activity Assessment: Participants' energy intake and expenditure, including dietary intake, as well as macronutrient, micronutrient, vitamin, and supplement intakes will be recorded at weeks 0 and 8 using a standardized Food Frequency and Activity Questionnaire (FFAQ). In addition, participants' nutrition knowledge will be assessed using the self-reported 97-item General and Sport-Specific Nutrition Knowledge Questionnaire (GeSNK) developed by Calella et al. (2017). The GeSNK encompasses 64 items assessing general and sport-specific nutrition knowledge, to explore knowledge regarding macro- and micronutrients in various food choices, awareness of diet-health associations, knowledge of fluid replacement, supplement intake, and food choices regarding sport recovery meals. As mentioned above, the GeSNK will be completed online along with the medical screening questions used to screen for inclusion criteria.

Sample size calculation

To our knowledge, no study has assessed the impact of dairy consumption on markers of bone metabolism and inflammation in male and female seniors. Using G*Power analysis for a repeated measures analysis of variance (3 intervention groups, 2 timepoints, sex as covariate), we calculated that a total sample size of n = 54 (i.e., 18 per intervention group) would be required to detect a medium effect of partial η2 = 0.06 with a power of (1-β) = 0.90, and a probability level of p = 0.05. Thus, the proposed total of 60 participants is more than adequate to detect significant effects and interactions, while allowing for a 20% attrition rate.

ELIGIBILITY:
Inclusion Criteria:

* Adults 55+ years from from the Niagara area.

Exclusion Criteria:

* injuries and inability to participate in classes,
* allergy to dairy foods/dairy protein, or
* diagnosed with lactose intolerance.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-08-10 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-08-28 (Actual)

PRIMARY OUTCOMES:
Serum concentrations of osteocalcin | Weeks 0 and 8
  Bone turnover marker measured in picograms/milliliter of serum (pg/mL)
Serum concentrations of amino-terminal propeptide of type I collagen (P1NP) | Weeks 0 and 8
  Bone formation marker measured in pg/mL
Serum concentrations of C-telopeptides of type I collagen (CTX) | Weeks 0 and 8
  Bone resorption marker measured in ng/mL
Serum concentrations of osteoprotegerin (OPG) | Weeks 0 and 8
  Regulator of bone remodelling (osteokine) measured in pg/mL
Serum concentrations of sclerostin | Weeks 0 and 8
  Regulator of bone remodelling (osteokine) measured in pg/mL
Serum concentrations of receptor activator of nuclear factor kappa-Β ligand (RANKL) | Weeks 0 and 8
  Regulator of bone remodelling (osteokine) measured in pg/mL
Serum concentrations of parathyroid hormone (PTH) | Weeks 0 and 8
  Regulator of bone remodelling measured in pg/mL
Plasma concentrations of interleukin-6 (IL6) | Weeks 0 and 8
  Inflammatory cytokine measured in pg/mL
Plasma concentrations of interleukin-10 (IL10) | Weeks 0 and 8
  Anti-inflammatory cytokine measured in pg/mL
plasma concentrations of inflammatory cytokines, including interleukin-6 (IL6), interleukin-10 Plasma concentrations of tumour necrosis factor-alpha (TNFα) | Weeks 0 and 8
  Pro-inflammatory cytokine measured in pg/mL
Serum concentrations of irisin | Weeks 0 and 8
  Myokine measured in pg/mL
Serum concentrations of insulin-like growth factor 1 (IGF1) | Weeks 0 and 8
  Growth factor measured in pg/mL

SECONDARY OUTCOMES:
Body mass | Weeks 0 and 8
  Body mass in kilograms (kg) using bioelectrical impedance analysis
Body composition | Weeks 0 and 8
  fat-free mass and fat mass in kg measured by bioelectrical impedance analysis
Height | Weeks 0 and 8
  Height measured in centimeters with a stadiometer
Energy intake and expenditure | Weeks 0 and 8
  Food Frequency and Activity Questionnaire
Sport-Specific Nutrition Knowledge Questionnaire (GeSNK) | Weeks 0 and 8
  A standardized questionnaire including 64 items assessing general and sport-specific nutrition knowledge.

CONTACTS AND LOCATIONS:
Locations (1):
- Brock University, St. Catharines, Ontario, Canada